CLINICAL TRIAL: NCT00088309
Title: Tenofovir Disoproxil Fumarate Salvage Therapy in HIV-Infected Children and a Study of Its Effect on Bone Metabolism
Brief Title: Effect of Tenofovir DF on Bone Metabolism in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040234; 04-C-0234
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-05

CONDITIONS: HIV Infections
Keywords: Drug Resistance; HAART; Pamidronate; Osteopenia; Pediatric; HIV; Pediatrics; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Bone Diseases, Metabolic | interventions — Diagnosis, Oral; Neuropsychological Tests

INTERVENTIONS:
Procedure: Eye exam
Procedure: Oral exam
Procedure: CT scan
Procedure: Neuropsychological testing
Procedure: Electrocardiogram
Procedure: Echocardiogram

SUMMARY:
This study will examine the long-term effects, particularly on bone metabolism, of the drug tenofovir DF in children with HIV infection. Tenofovir DF is approved for treating HIV-infected adults, but its use in children has not yet been approved. The drug may be helpful for children who have been treated with many other drugs and still have detectable HIV in their blood despite ongoing therapy. In a previous study, many children given tenofovir DF responded well, with increases in T-cell counts and decreases in viral load. However, many children also experienced bone thinning. This study will explore the problem of bone thinning in children taking tenofovir DF in combination with highly active antiretroviral therapy (HAART).

HIV-infected patients from 4 to 20 years old who are taking tenofovir DF or for whom tenofovir DF treatment has been recommended may be eligible for this 3-year study.

Participants take tenofovir DF every day in addition to their antiretroviral therapy. They have frequent follow-up visits for tests and procedures as follows:

* Study days 0, 2, and 4: blood tests.
* Screening and every study visit starting day 6: Physical exam, medical history, blood and urine tests.
* Baseline and every 48 weeks: Dental and eye examinations, kidney ultrasound, tuberculin skin testing, chest x-ray, electrocardiogram and echocardiogram, computed tomography (CT) scan, neuropsychological testing and neurologic assessment.
* The bone age hand x-rays are done every 24 weeks, unless the growth plates are fused (i.e. the child has stopped growing)
* DEXAs are done at 0, 12, 24 weeks and every 24 weeks thereafter. Dual energy x-ray absorptionometry (DEXA) scan is used to assess bone density. The patient lies still on a table while the spine and hip are scanned using a small amount of radiation. Only the spine and hip are scanned in the DEXA scan test.
* Baseline and week 24: Optional bone biopsy. Some patients are asked to undergo a bone biopsy to better understand the effect of Tenofovir DF on bone. For the procedure, the child is given a sedative. The skin over the hipbone is numbed with a small needle, a small incision is made and a larger needle is inserted into the bone. Some of the bone tissue is withdrawn through the needle and the incision is closed.
* Possible lumbar puncture (spinal tap): This optional procedure analyzes cerebrospinal fluid (CSF), the fluid that bathes the brain and spinal cord. The patient is given a local anesthetic and a needle is inserted into the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle. There is no specific schedule for this procedure if the patient opts for it.

Patients who are benefiting from tenofovir DF therapy but show signs of bone effects are offered treatment with pamidronate (Aredia), a drug used to treat hypercalcemia (too much calcium in the blood). Patients who stop taking tenofovir DF because of bone toxicity continue to be followed on the regular study schedule. Those who stop the drug for toxicity other than bone toxicity or for toxicity not related to tenofovir DF are followed every 4 weeks until their laboratory test results improve.

DETAILED DESCRIPTION:
Tenofovir disoproxil fumarate (TDF) was approved for the treatment of HIV-infected adults in October 2001. In November 2001, we began enrollment to our phase I/II study of tenofovir DF in HIV-infected children (02-C-0006). That study has completed enrollment. The virologic and immunologic responses seen on that study in a group of heavily treatment-experienced children with multidrug resistant HIV were surprisingly good. The drug was well tolerated, but significant decreases in bone mineral density were seen in a minority of patients.

With the current study we will enroll and systematically investigate HIV-infected children for whom tenofovir DF is being used as part of salvage combination HIV therapy. The primary objective of the study is to characterize the change in bone mineral density (BMD), as measured by lumbar spine dual-energy x-ray absorptiometry (DEXA), during and following treatment with tenofovir DF-containing antiretroviral therapy in HIV-infected children. The study will enroll 3 cohorts of children: 1) HIV-infected children about to start a tenofovir DF-containing antiretroviral regimen, 2) HIV-infected children already on tenofovir DF with available baseline DEXA results, and 3) HIV-infected children already on tenofovir DF but without baseline DEXA results who will come here for investigations of bone metabolism. Studies of bone metabolism will include periodic measurements of serum and urine calcium and phosphorus, PTH and vitamin D levels, bone resorption markers (urinary collagen cross-linked N-telopeptide and free deoxypyridinoline), bone formation markers (serum osteocalcin and bone specific alkaline phosphatase), IGF-1 levels, bone age, and DEXA scans. Patients about to start tenofovir DF (cohort 1) will be offered the option of having a transiliac crest core bone biopsy with tetracycline labeling performed at baseline and at 6 months to assess static and dynamic parameters of bone quality and turnover (histomorphometry). Subjects with substantial presumed tenofovir DF-related bone toxicity who are deriving benefit from their tenofovir DF-containing antiretroviral drug regimen will be offered the option of pamidronate therapy. The effects of pamidronate treatment on bone toxicity associated with tenofovir DF in these patients will be assessed in an exploratory fashion. It is expected that up to 40 patients with baseline BMD measurements will be enrolled onto this protocol. An additional 10 patients who are undergoing tenofovir DF treatment but who did not receive baseline BMD measurements will also be permitted to enroll in order to contribute to the data used to characterize changes in toxicity.

ELIGIBILITY:
INCLUSION CRITERIA: Cohort 1 - patients about to start tenofovir DF

* HIV-infected children between the ages of 4 years and less than 21 years.
* Clinical decision has been made to start the patient on tenofovir DF-containing antiretroviral regimen
* BSA greater than or equal to 0.85 m2
* Sexually active patients must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.
* Not pregnant or breast feeding
* 25-OH-Vitamin D level greater than 20 ng/ml (supplementation allowed)
* Less than or equal to grade 1 serum calcium or ionized calcium (supplementation allowed)
* AST and ALT less than or equal to 7.5 times the upper limit of normal
* Age-adjusted normal serum creatinine OR a creatinine clearance greater than or equal to 70 mL/min/1.73.
* Informed consent: patient, parent or legal guardian must sign the study informed consent to document their understanding of the investigational nature and the risks of the study before any protocol-related studies are performed.

INCLUSION CRITERIA: Cohort 2 - patients already being treated with tenofovir DF who have baseline DEXA available

* HIV-infected children between the ages of 4 years and less than 21 years.
* Current tenofovir DF-containing antiretroviral regimen was started less than 6 months ago
* Baseline DEXA for L-spine BMD is available and was performed less than six months prior to or within the first week of starting tenofovir DF
* BSA greater than or equal to 0.85 m2
* Sexually active patients must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.
* Not pregnant or breast feeding
* 25-OH-Vitamin D level greater than 20 ng/ml (supplementation allowed)
* Less than or equal to grade 1 serum calcium or ionized calcium (supplementation allowed)
* AST and ALT less than or equal to 7.5 times the upper limit of normal
* Age-adjusted normal serum creatinine OR a creatinine clearance greater than or equal to 70 mL/min/1.73.
* Informed consent: patient, parent or legal guardian must sign the study informed consent to document their understanding of the investigational nature and the risks of the study before any protocol-related studies are performed.

INCLUSION CRITERIA: Cohort 3 - patients already being treated with an antiretroviral regimen that includes tenofovir DF who DO NOT have baseline DEXA available

* HIV-infected children between the ages of 4 years and less than 21 years.
* Current antiretroviral regimen includes tenofovir DF
* Baseline (within prior 6 months) DEXA for L-spine BMD is NOT available
* BSA greater than or equal to 0.85 m2
* Sexually active patients must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.
* Not pregnant or breast feeding
* 25-OH-Vitamin D level greater than 20 ng/ml (supplementation allowed)
* less than or equal to grade 1 serum calcium or ionized calcium (supplementation allowed)
* AST and ALT less than or equal to 7.5 times the upper limit of normal
* Age-adjusted normal serum creatinine (see table below) OR a creatinine clearance greater than or equal to 70 mL/min/1.73.
* Informed consent: patient, parent or legal guardian must sign the study informed consent to document their understanding of the investigational nature and the risks of the study before any protocol-related studies are performed.

INCLUSION CRITERIA: Eligibility criteria for pamidronate therapy (after enrollment on protocol)

One of the following while on tenofovirDF-containing antiretroviral regimen:

* Greater than 6% loss in L-spine BMD in the presence of a BMD Z score less than -2.5 at 6 months compared to baseline
* Minimal trauma fracture
* BMD Z-score less than -3

AND

One of the following while on tenofovirDF-containing antiretroviral regimen:

* Greater than or equal to 0.5 log decrease in VL from baseline
* Greater than or equal to 25% increase in absolute CD4 count from baseline

Improvement in HIV-related signs or symptoms

OR

BMD Z-score less than -3 (i.e., pamidronate therapy will also be considered for subjects whose BMD Z score is less than -3 at baseline)

* Age-adjusted normal serum creatinine (see table below) OR a creatinine clearance greater than or equal to 70 mL/min/1.73.
* Less than or equal to grade 1 serum phosphate, magnesium, and potassium (supplementation allowed)
* Not pregnant or breast feeding
* No history of hypersensitivity to bisphosphonates

INCLUSION CRITERIA: Eligibility criteria for bone biopsy (after enrollment on protocol)

* No history of bleeding abnormality
* No history of hypersensitivity or intolerance to tetracycline or related drugs
* Normal CBC and PT/PTT
* BMD Z-score greater than -3
* Informed consent: patient, parent or legal guardian must sign a separate informed consent to document their understanding of the investigational nature and the risks of the bone biopsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2004-06; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sleasman JW, Nelson RP, Goodenow MM, Wilfret D, Hutson A, Baseler M, Zuckerman J, Pizzo PA, Mueller BU. Immunoreconstitution after ritonavir therapy in children with human immunodeficiency virus infection involves multiple lymphocyte lineages. J Pediatr. 1999 May;134(5):597-606. doi: 10.1016/s0022-3476(99)70247-7. PMID 10228296
- [Background] Gortmaker SL, Hughes M, Cervia J, Brady M, Johnson GM, Seage GR 3rd, Song LY, Dankner WM, Oleske JM; Pediatric AIDS Clinical Trials Group Protocol 219 Team. Effect of combination therapy including protease inhibitors on mortality among children and adolescents infected with HIV-1. N Engl J Med. 2001 Nov 22;345(21):1522-8. doi: 10.1056/NEJMoa011157. PMID 11794218
- [Background] Wainberg MA, Miller MD, Quan Y, Salomon H, Mulato AS, Lamy PD, Margot NA, Anton KE, Cherrington JM. In vitro selection and characterization of HIV-1 with reduced susceptibility to PMPA. Antivir Ther. 1999;4(2):87-94. doi: 10.1177/135965359900400205. PMID 10682153